CLINICAL TRIAL: NCT06886958
Title: Spectral CT Protocol Optimization for Atherosclerotic Plaque CharacterizatION
Acronym: SCORPION
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS SYNLAB SDN (Other)
Collaborators: Fondazione Monasterio/CNR (Unknown)
Responsible Party: Sponsor
Other Study IDs: 7/22
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Atherosclerotic Disease
Keywords: Atherosclerotic Plaque; Dual-Energy CT (DECT); Photon-Counting CT (PCCT); Radiomics; Cardiovascular Risk Stratification
MeSH Terms: conditions — Plaque, Atherosclerotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cardiovascular Imaging patiets: Patients who have undergone DECT for cardiovascular imaging (coronary and/or carotid) or with critical stenosis

SUMMARY:
The SCORPION study (Spectral CT Protocol Optimization for Atherosclerotic Plaque Characterization) is a retrospective and prospective observational research project aimed at improving the diagnostic accuracy of dual-energy CT (DECT) and photon-counting CT (PCCT) in the characterization of atherosclerotic plaques in the coronary and carotid arteries. Given that cardiovascular diseases remain a leading cause of mortality despite advances in prevention and treatment, optimizing non-invasive imaging methods is crucial. CT Angiography (CTA) has become the gold standard for diagnosing coronary artery disease and carotid stenosis, but existing techniques require enhancement to improve plaque characterization, which is vital for risk stratification and patient management. While DECT has demonstrated potential in differentiating tissue types, its clinical adoption has been slow due to a lack of broad validation. This study seeks to establish a standardized imaging protocol that will provide more precise and reproducible plaque characterization.

The primary objective of the study is to develop a standardized method for characterizing atherosclerotic plaques using DECT based on retrospective datasets from Synlab. The first secondary objective is to validate this workflow with photon-counting CT data from an independent cohort at Fondazione Monasterio/CNR, ensuring the reliability of the technique across different imaging modalities. The second secondary objective involves defining an optimized DECT protocol using the energy spectrum of PCCT, ultimately refining imaging parameters for improved plaque assessment.

The study is structured into two phases. In the retrospective phase, data from fifty patients with critical stenosis (greater than 75% narrowing of the artery) who previously underwent DECT scans are analyzed. This step focuses on optimizing imaging parameters, segmentation techniques, and post-processing workflows. In the prospective phase, another cohort of fifty patients undergoes scanning with photon-counting CT to validate the workflow developed in the first phase. The results will inform the refinement of an optimized DECT protocol, translating the benefits of photon-counting technology into more widely available DECT scanners.

Patients included in the study must be at least sixty years old and have undergone DECT for cardiovascular imaging of the coronary or carotid arteries. The imaging process involves a third-generation dual-energy CT scanner (Somatom Force, Siemens) with high-resolution imaging settings, dual-energy tube voltages of 150 and 90 kV, ECG-gated acquisition, and the use of iodine contrast. The collected data is processed using various reconstruction techniques to extract quantitative imaging biomarkers, including total plaque volume, non-calcified and calcified plaque volumes, remodeling index, and degree of luminal stenosis. The study employs PyRadiomics, an open-source platform for radiomic feature extraction, to standardize data analysis and improve reproducibility.

The expected outcome of this research is an improved molecular characterization of atherosclerosis, leading to more accurate risk stratification and predictive models for cardiovascular events. By refining imaging techniques, the study aims to enhance diagnostic precision and minimize unnecessary hospitalizations, ultimately improving patient outcomes. Furthermore, establishing a standardized DECT protocol will allow for broader clinical adoption, making advanced plaque characterization more accessible in routine cardiovascular assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone DECT for cardiovascular imaging (coronary and/or carotid)
* Patients with critical stenosis (>75% diameter, coronary or carotid artery) aged > 60aa

Exclusion Criteria:

* Patients negative for critical stenosis (<75% diameter) and/or imaging artefacts (e.g. due to movement, swallowing, or arrhythmias).
* Patients under 60 years of age
* Patients allergic to iodinated contrast medium (prospective phase)
* Patients with chronic renal insufficiency (prospective phase)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects over 60 years of age performing a cardiovascular imaging examination
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Imaging analyses | 1 - 24 months
  Extraction of numerical data from imaging for the generation of a reproducible and standardized method for characterising the various components of atherosclerotic plaques

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Cavaliere, MD, Principal Investigator — carlo.cavaliere@synlab.it
Locations (1):
- Laura Pierri, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Griethuysen JJM, Fedorov A, Parmar C, Hosny A, Aucoin N, Narayan V, Beets-Tan RGH, Fillion-Robin JC, Pieper S, Aerts HJWL. Computational Radiomics System to Decode the Radiographic Phenotype. Cancer Res. 2017 Nov 1;77(21):e104-e107. doi: 10.1158/0008-5472.CAN-17-0339. PMID 29092951
- [Background] Forghani R, De Man B, Gupta R. Dual-Energy Computed Tomography: Physical Principles, Approaches to Scanning, Usage, and Implementation: Part 1. Neuroimaging Clin N Am. 2017 Aug;27(3):371-384. doi: 10.1016/j.nic.2017.03.002. PMID 28711199
- [Background] Yeboah J, McClelland RL, Polonsky TS, Burke GL, Sibley CT, O'Leary D, Carr JJ, Goff DC, Greenland P, Herrington DM. Comparison of novel risk markers for improvement in cardiovascular risk assessment in intermediate-risk individuals. JAMA. 2012 Aug 22;308(8):788-95. doi: 10.1001/jama.2012.9624. PMID 22910756
- [Background] Erbel R, Mohlenkamp S, Moebus S, Schmermund A, Lehmann N, Stang A, Dragano N, Gronemeyer D, Seibel R, Kalsch H, Brocker-Preuss M, Mann K, Siegrist J, Jockel KH; Heinz Nixdorf Recall Study Investigative Group. Coronary risk stratification, discrimination, and reclassification improvement based on quantification of subclinical coronary atherosclerosis: the Heinz Nixdorf Recall study. J Am Coll Cardiol. 2010 Oct 19;56(17):1397-406. doi: 10.1016/j.jacc.2010.06.030. PMID 20946997
- [Background] Yamak D, Panse P, Pavlicek W, Boltz T, Akay M. Non-calcified coronary atherosclerotic plaque characterization by dual energy computed tomography. IEEE J Biomed Health Inform. 2014 May;18(3):939-45. doi: 10.1109/JBHI.2013.2295534. PMID 24808227
- [Background] Mandal SR, Bharati A, Haghighi RR, Arava S, Ray R, Jagia P, Sharma S, Chatterjee S, Tabin M, Sharma M, Sharma S, Kumar P. Non-invasive characterization of coronary artery atherosclerotic plaque using dual energy CT: Explanation in ex-vivo samples. Phys Med. 2018 Jan;45:52-58. doi: 10.1016/j.ejmp.2017.12.006. Epub 2017 Dec 19. PMID 29472090
- [Background] Haghighi RR, Chatterjee S, Tabin M, Sharma S, Jagia P, Ray R, Singh RP, Yadav R, Sharma M, Krishna K, Vani VC, Lakshmi R, Mandal SR, Kumar P, Arava S. DECT evaluation of noncalcified coronary artery plaque. Med Phys. 2015 Oct;42(10):5945-54. doi: 10.1118/1.4929935. PMID 26429269
- [Background] Obaid DR, Calvert PA, Gopalan D, Parker RA, West NE, Goddard M, Rudd JH, Bennett MR. Dual-energy computed tomography imaging to determine atherosclerotic plaque composition: a prospective study with tissue validation. J Cardiovasc Comput Tomogr. 2014 May-Jun;8(3):230-7. doi: 10.1016/j.jcct.2014.04.007. Epub 2014 May 2. PMID 24939072
- [Background] Tanami Y, Ikeda E, Jinzaki M, Satoh K, Nishiwaki Y, Yamada M, Okada Y, Kuribayashi S. Computed tomographic attenuation value of coronary atherosclerotic plaques with different tube voltage: an ex vivo study. J Comput Assist Tomogr. 2010 Jan;34(1):58-63. doi: 10.1097/RCT.0b013e3181b66c41. PMID 20118723
- [Background] Barreto M, Schoenhagen P, Nair A, Amatangelo S, Milite M, Obuchowski NA, Lieber ML, Halliburton SS. Potential of dual-energy computed tomography to characterize atherosclerotic plaque: ex vivo assessment of human coronary arteries in comparison to histology. J Cardiovasc Comput Tomogr. 2008 Jul-Aug;2(4):234-42. doi: 10.1016/j.jcct.2008.05.146. Epub 2008 Jun 12. PMID 19083956
- [Background] Narula J, Nakano M, Virmani R, Kolodgie FD, Petersen R, Newcomb R, Malik S, Fuster V, Finn AV. Histopathologic characteristics of atherosclerotic coronary disease and implications of the findings for the invasive and noninvasive detection of vulnerable plaques. J Am Coll Cardiol. 2013 Mar 12;61(10):1041-51. doi: 10.1016/j.jacc.2012.10.054. PMID 23473409
- [Background] Kalisz K, Halliburton S, Abbara S, Leipsic JA, Albrecht MH, Schoepf UJ, Rajiah P. Update on Cardiovascular Applications of Multienergy CT. Radiographics. 2017 Nov-Dec;37(7):1955-1974. doi: 10.1148/rg.2017170100. PMID 29131773
- [Background] Cademartiri F, Seitun S, Clemente A, La Grutta L, Toia P, Runza G, Midiri M, Maffei E. Myocardial blood flow quantification for evaluation of coronary artery disease by computed tomography. Cardiovasc Diagn Ther. 2017 Apr;7(2):129-150. doi: 10.21037/cdt.2017.03.22. PMID 28540209
- [Background] Johnson TR, Krauss B, Sedlmair M, Grasruck M, Bruder H, Morhard D, Fink C, Weckbach S, Lenhard M, Schmidt B, Flohr T, Reiser MF, Becker CR. Material differentiation by dual energy CT: initial experience. Eur Radiol. 2007 Jun;17(6):1510-7. doi: 10.1007/s00330-006-0517-6. Epub 2006 Dec 7. PMID 17151859
- [Background] Puchner SB, Liu T, Mayrhofer T, Truong QA, Lee H, Fleg JL, Nagurney JT, Udelson JE, Hoffmann U, Ferencik M. High-risk plaque detected on coronary CT angiography predicts acute coronary syndromes independent of significant stenosis in acute chest pain: results from the ROMICAT-II trial. J Am Coll Cardiol. 2014 Aug 19;64(7):684-92. doi: 10.1016/j.jacc.2014.05.039. PMID 25125300
- [Background] Motoyama S, Sarai M, Harigaya H, Anno H, Inoue K, Hara T, Naruse H, Ishii J, Hishida H, Wong ND, Virmani R, Kondo T, Ozaki Y, Narula J. Computed tomographic angiography characteristics of atherosclerotic plaques subsequently resulting in acute coronary syndrome. J Am Coll Cardiol. 2009 Jun 30;54(1):49-57. doi: 10.1016/j.jacc.2009.02.068. PMID 19555840
- [Background] Grundy SM, Stone NJ. 2018 American Heart Association/American College of Cardiology/Multisociety Guideline on the Management of Blood Cholesterol-Secondary Prevention. JAMA Cardiol. 2019 Jun 1;4(6):589-591. doi: 10.1001/jamacardio.2019.0911. No abstract available. PMID 30994869